CLINICAL TRIAL: NCT06030271
Title: A Prospective, Non-Randomized Pivotal Clinical Investigation to Demonstrate the Safety and Performance of the TrueCross Single-Use Microcatheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insight Lifetech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-003C
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease Obliterative; Chronic Total Occlusion (CTO)
Keywords: microcatheter, CTO, coronary artery disease, PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TrueCross microcatheter (Experimental): The TrueCross Single-use Microcatheter will be used in percutaneous coronary intervention(PCI) of the enrolled subjects.
  Interventions: Device: Microcatheter

INTERVENTIONS:
Device: Microcatheter — Support and facilitate the placement of the guidewire in the coronary artery with a CTO.
  Other Names: TrueCross

SUMMARY:
The trial is a pivotal clinical investigation, which is a prospective, non-randomized pivotal clinical investigation to demonstrate the safety and performance of the TrueCross Single-use Microcatheter.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate the performance and safety of the TrueCross Single-use Microcatheter in patients requiring a PCI procedure as well as the related clinical benefits.

The study will include 59 subjects suffering from coronary artery disease requiring a percutaneous coronary intervention. Enrollment duration will be 4 months or so without follow-up. It is a single-arm trial.In the uneventual case of a potential dropout (serious protocol deviation or procedure interruption unrelated to the catheter), subjects will be replaced to reach 59 evaluable subjects for the Per Protocol population.

ELIGIBILITY:
Inclusion Criteria:

i. Subjects who are >25 years of age. ii. Subjects who are able/willing to provide a written informed consent prior to participating in the clinical investigation.

iii. The subject is male or, if female, is either not of childbearing potential or must use effective contraception during participation in this Clinical Investigation.

iv. Subject suffering from coronary artery disease requiring percutaneous coronary angiography and/or intervention.

v. Lesions classified as CTOs, meaning, TIMI 0 flow within the occluded segment and angiographic or clinical evidence or high likelihood of an occlusion duration > 3 months vi. Reference vessel diameter ≥2 mm.

Exclusion Criteria:

i. Coronary angiography and/or intervention contraindications. ii. Subjects with severe arrhythmia. iii. Subjects with severe systemic infection. iv. Subjects with severe coagulation disorder. v. Subjects with severe heart failure, unstable decompensated heart failure, congestive heart failure, or dyspnea who are unable to lie supine on the examination table for angiography.

vi. Subjects with prior coronary artery spams or prior heart valve replacement. vii. Currently participating in an investigational drug or another device clinical investigation that has not completed the primary endpoint or that clinically interferes with the current clinical investigation endpoints.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical Performance-technical success | during the procedure
  Angiographic confirmation of the TrueCross Single-use Microcatheter's ability to support the guidewire in crossing the CTO in the target vessel true lumen.

SECONDARY OUTCOMES:
Safety-observation of AE | ADE: during the procedure; non-device/procedure related AE: from screening start to the end of the procedure
  Occurrence of any device related adverse event during use of the microcatheter throughout the procedure.
  Occurrence of any non-device/procedure related events from screening start to the end of the procedure. This will include any events related or cause by other devices used independently from the TrueCross Single-use Microcatheter during the same PCI procedure.
Clinical Performance/Effectiveness | during the procedure
  1. Angiographic confirmation of successful placement and successful injection of contrast medium into the vessel lumen,
  2. Ability of exchange of the guidewire,
  3. Safe withdrawal of the TrueCross Single-use Microcatheter.
  4. Procedural efficiency measures (procedure time and injected contrast volume).

CONTACTS AND LOCATIONS:
Locations (7):
- Georgia (4):
  - Israeli-Georgian Medical Research Clinic Ltd - Healthycore Clinic, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - Tbilisi Institute of Medicine, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
- Greece (2):
  - Onassis Heart Surgery Centre, Athens
  - Red Cross General Hospital, Athens
- National Heart Centre Singapore, Singapore, Singapore